CLINICAL TRIAL: NCT01949584
Title: Study of Nasal Airflow Pressure Optimization to Resolve Excessive Snoring
Acronym: SNORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: inSleep Technologies, LLC (Industry)
Collaborators: Johns Hopkins University (Other); Doctors Community Hospital (Unknown); NeuroTrials Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IS103-PRO-00002
Record Dates: First submitted 2013-09-20; First posted 2013-09-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Snoring
MeSH Terms: conditions — Snoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: nasal continuous positive airway pressure less than or equal to 6 cm H2O — Low level continuous positive airway pressure delivered during sleep.
  Other Names: Cloud9™ nasal CPAP device and nasal interface

SUMMARY:
This is a prospective, interventional, study in which patients with a history of habitual snoring to determine whether low pressure nasal continuous airway pressure can reduce the frequency, duration or intensity of snoring in subjects with mild to moderate snoring who do not have Obstructive Sleep Apnea (OSA).

DETAILED DESCRIPTION:
In this a prospective, interventional, study, each patient will be studied four times. Subjects without OSA will undergo an initial observational control study to establish the presence of snoring (session 1); a single CPAP titration night to determine the minimally effective CPAP level (session 2) to alleviate snoring; a subsequent full night of CPAP treatment at this CPAP level (CPAP not to exceed 6 cm H2O) using the Cloud9™ low-pressure CPAP device (session 3); and a final control night of study conducted off CPAP to assess whether the patient's snoring remained stable over time (session 4). In this study, each subject shall serve as his/her own control.

ELIGIBILITY:
Inclusion Criteria:

* Subject is > 18 years of age.
* Subject is willing and able to provide written Informed Consent using a Patient Information and Consent form that has been reviewed and approved by a governing Institutional Review Board (IRB).
* Subject has a history of habitual snoring (almost every night or every night for at least 30% of the night) as determined by the subject or a bed-partner.
* Subject has been pre-screened and demonstrates no excess daytime sleepiness on an Epworth Questionnaire (an assessment of daytime sleepiness; high number = greater sleepiness) score of less than 11, no history of witnessed apneas or nocturnal gasping/choking episodes and a body mass index (BMI) ≤ 35.

Inclusion Criteria for treatment trials (Nights 2 and 3):

* Subject meets Inclusion Criteria for the Baseline Trial (criteria a-d above)
* The subject has snoring intensity that exceeds 40 dBA during ≥30% of the respiratory efforts during sleep time on the baseline study night.

Exclusion Criteria:

* Subject has been diagnosed with COPD (Chronic Obstructive Pulmonary Disease), such as asthma, emphysema or chronic bronchitis.
* Subject has a history of heart disease, heart attack or stroke.
* Subject has uncontrolled or poorly controlled hypertension.
* Subject has been diagnosed with Obstructive Sleep Apnea (OSA), defined as an apnea hypopnea index (AHI) ≥ 5/hr in the presence of excessive sleepiness (an Epworth score ≥ 11) or AHI ≥15/hr when there is no evidence of excessive daytime sleepiness (an Epworth score ≤ 10).
* Subject is currently participating in another clinical study for which follow-up is ongoing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-08; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Efficacy - The Cloud9™ device is expected to reduce the incidence of snoring. | single night of sleep
  The primary objective of this study is to demonstrate that minimally effective nasal CPAP (≤ 6 cm H2O) delivered by the Cloud9™ device reduces the number of snoring events and reduces snoring intensity in habitual, simple snorers in treatment session 3. We will test the hypothesis that the Cloud9™ device will decrease the number of loud snores by 50% or decrease the overall number of snores by 50%.

SECONDARY OUTCOMES:
Safety - Adverse events associated with CPAP (nasal or skin irritation, epistaxis and sleep disruption) will occur in few subjects. | two different single nights
  Safety- Adverse events associated with the Cloud9™ device (nasal or skin irritation, epistaxis and sleep disruption) will occur in fewer than 20% of the subjects in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lauk, Study Director — inSleep Tech
Locations (3):
- United States (3):
  - NeuroTrials Research, Inc., Atlanta, Georgia
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Doctors Community Hospital, Lanham, Maryland

REFERENCES:
- [Derived] Guzman MA, Sgambati FP, Pho H, Arias RS, Hawks EM, Wolfe EM, Otvos T, Rosenberg R, Dakheel R, Schneider H, Kirkness JP, Smith PL, Schwartz AR. The Efficacy of Low-Level Continuous Positive Airway Pressure for the Treatment of Snoring. J Clin Sleep Med. 2017 May 15;13(5):703-711. doi: 10.5664/jcsm.6588. PMID 28356182